CLINICAL TRIAL: NCT01413204
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter Study to Evaluate the Efficacy, Safety, and Tolerability of TA-7284 as Monotherapy in the Treatment of Subjects With Type 2 Diabetes Mellitus
Brief Title: Efficacy and Safety Study of TA-7284 in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TA-7284-05
Record Dates: First submitted 2011-08-04; First posted 2011-08-10 (Estimated); Results first posted 2014-06-05 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: TA-7284; JNJ-28431754; Canagliflozin; Sodium Glucose Co-transporter (SGLT2 inhibitor)
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- TA-7284 Low (Experimental)
  Interventions: Drug: TA-7284 Low
- TA-7284 High (Experimental)
  Interventions: Drug: TA-7284 High
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TA-7284 Low — The patients will receive TA-7284-Low orally for 24 weeks.
  Arms: TA-7284 Low
Drug: TA-7284 High — The patients will receive TA-7284-High orally for 24 weeks.
  Arms: TA-7284 High
Drug: Placebo — The patients will receive Placebo orally for 24 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of TA-7284 as monotherapy in patients with type 2 Diabetes for 24 weeks administration.

DETAILED DESCRIPTION:
This is a randomized, 3-arm, parallel group, double blind study to evaluate the efficacy and safety of TA-7284 in Japanese patients with Type 2 diabetes mellitus, who are not optimally controlled on diet and exercise. The patients will receive either TA-7284-Low, TA-7284-High or Placebo orally alone for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Men or women age ≥20 years old
* Diagnosed with Type 2 diabetes mellitus at least 3 months before run-in period
* HbA1c of ≥7.0% and ≤10.0%

Exclusion Criteria:

* Type I diabetes mellitus, diabetes mellitus resulting from pancreatic disorder, secondary diabetes mellitus
* Past or current history of severe diabetic complications
* Fasting plasma glucose > 270 mg/dL before treatment start
* History of hereditary glucose-galactose malabsorption or primary renal glucosuria
* Patients requiring insulin therapy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2011-07; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nobuya Inagaki, M.D., Study Director — Kyoto University, Graduate School of Medicine; Kazuoki Kondo, M.D., Study Director — Tanabe Pharma Corporation
Locations (5):
- Japan (5):
  - Reserch site, Chūbu
  - Reserch site, Kanto
  - Reserch site, Kinki
  - Reserch site, Shikoku
  - Reserch site, Tōhoku

REFERENCES:
- [Derived] Inagaki N, Kondo K, Yoshinari T, Takahashi N, Susuta Y, Kuki H. Efficacy and safety of canagliflozin monotherapy in Japanese patients with type 2 diabetes inadequately controlled with diet and exercise: a 24-week, randomized, double-blind, placebo-controlled, Phase III study. Expert Opin Pharmacother. 2014 Aug;15(11):1501-15. doi: 10.1517/14656566.2014.935764. PMID 25010793

RESULTS

PARTICIPANT FLOW:
Groups:
- TA-7284 Low: TA-7284 low dose, once daily for 24 weeks
- TA-7284 High: TA-7284 high dose, once daily for 24 weeks
- Placebo: TA-7284 Placebo, once daily for 24 weeks
Period: Overall Study
Arm/Group | TA-7284 Low | TA-7284 High | Placebo
Started | 90 | 89 | 93
Completed | 84 | 83 | 74
Not Completed | 6 | 6 | 19
Not completed — Adverse Event | 1 | 2 | 2
Not completed — Physician Decision | 3 | 0 | 2
Not completed — Withdrawal by Subject | 1 | 4 | 4
Not completed — Clearly not eligible for the study | 0 | 0 | 1
Not completed — Fasting plasma glucose level increased | 1 | 0 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TA-7284 Low | TA-7284 High | Placebo | Total
Number analyzed (Participants) | 90 | 89 | 93 | 272
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (10.4) | 57.3 (11.1) | 58.2 (11) | 58 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 16 | 33 | 80
  Male | 59 | 73 | 60 | 192

OUTCOME MEASURES:

1. Primary Outcome: Change in Hemoglobin A1c (A1C) From Baseline (NGSP Value)
Time Frame: baseline and 24 weeks
Population: Full analysis set, last observation carried forward
Measure: Least Squares Mean (Standard Error); unit: percent HbA1C
Arm/Group | TA-7284 Low | TA-7284 High | Placebo
Number analyzed (Participants) | 90 | 88 | 93
percent HbA1C | -0.74 (0.07) | -0.76 (0.07) | 0.29 (0.07)

2. Secondary Outcome: Change in Fasting Plasma Glucose
Time Frame: Week 24
Reporting Status: Not Posted

3. Secondary Outcome: Change in Body Weight
Time Frame: Week 24
Reporting Status: Not Posted

4. Secondary Outcome: Change in Blood Pressure
Time Frame: Week 24
Reporting Status: Not Posted

5. Secondary Outcome: Change in Postprandial Plasma Glucose, Insulin and Urinary Glucose Excretion After a 75 g Oral Glucose Tolerance Test
Time Frame: Week 24
Reporting Status: Not Posted

6. Secondary Outcome: Safety and Tolerability Assessed by Adverse Events, Hypoglycemic Events, Laboratory Tests, 12-lead ECG and Vital Signs
Time Frame: Week 24
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 26 weeks
Arm/Group | TA-7284 Low | TA-7284 High | Placebo
Serious Adverse Events (participants affected / at risk) | 1/90 | 1/89 | 2/93
Other Adverse Events (participants affected / at risk) | 59/90 | 55/89 | 54/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TA-7284 Low (N=90) | TA-7284 High (N=89) | Placebo (N=93)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Oropharyngeal cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TA-7284 Low (N=90) | TA-7284 High (N=89) | Placebo (N=93)
Abdominal discomfort (Gastrointestinal disorders) | 3 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Acute tonsillitis (Infections and infestations) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Asteatosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1
Bacteriuria (Infections and infestations) | 1 | 0 | 0
Balanoposthitis (Reproductive system and breast disorders) | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 2
Blood creatinine increased (Investigations) | 1 | 0 | 0
Blood ketone body increased (Investigations) | 3 | 7 | 2
Blood parathyroid hormone increased (Investigations) | 0 | 1 | 0
Blood pressure increased (Investigations) | 0 | 2 | 4
Blood triglycerides increased (Investigations) | 0 | 0 | 2
Blood uric acid increased (Investigations) | 0 | 0 | 1
Blood urine present (Investigations) | 3 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 1 | 0
Cervicobrachial syndrome (Nervous system disorders) | 1 | 0 | 0
Chest discomfort (General disorders) | 1 | 0 | 0
Chronic sinusitis (Infections and infestations) | 1 | 0 | 0
Colonic polyp (Gastrointestinal disorders) | 0 | 0 | 1
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 4 | 1
Contusion (Injury, poisoning and procedural complications) | 2 | 4 | 2
Cystitis (Infections and infestations) | 0 | 1 | 1
Dental caries (Gastrointestinal disorders) | 2 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0
Diplopia (Eye disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1
Dizziness postural (Nervous system disorders) | 1 | 0 | 1
Dry eye (Eye disorders) | 1 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 3 | 1
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 1 | 2
Enteritis infectious (Infections and infestations) | 0 | 1 | 1
Enterocolitis (Gastrointestinal disorders) | 2 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Face injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Folliculitis (Infections and infestations) | 1 | 1 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 2 | 1 | 3
Gastritis atrophic (Gastrointestinal disorders) | 1 | 1 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 1
Gingivitis (Gastrointestinal disorders) | 2 | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Hangover (General disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 1 | 0
Heat rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 1
Herpes virus infection (Infections and infestations) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0
Hordeolum (Infections and infestations) | 1 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0
Hunger (General disorders) | 1 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 3
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 1 | 2
Hypoglycaemia unawareness (Metabolism and nutrition disorders) | 4 | 5 | 2
Influenza (Infections and infestations) | 3 | 0 | 2
Injury corneal (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 2 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Migraine (Nervous system disorders) | 0 | 1 | 0
Mouth injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 19 | 16 | 27
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Nephropathy (Renal and urinary disorders) | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Palpitations (Cardiac disorders) | 1 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
Periodontal disease (Gastrointestinal disorders) | 0 | 1 | 1
Periodontitis (Gastrointestinal disorders) | 3 | 3 | 1
Pharyngitis (Infections and infestations) | 6 | 1 | 1
Pharyngitis bacterial (Infections and infestations) | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 4 | 1 | 1
Polycythaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Post herpetic neuralgia (Nervous system disorders) | 0 | 1 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulpitis dental (Infections and infestations) | 0 | 2 | 1
Punctate keratitis (Eye disorders) | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Sciatica (Nervous system disorders) | 0 | 1 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skeletal injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0
Thirst (General disorders) | 0 | 0 | 1
Tinea pedis (Infections and infestations) | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0
Urine albumin/creatinine ratio increased (Investigations) | 0 | 1 | 1
Urine ketone body present (Investigations) | 1 | 3 | 0
Urine output increased (Investigations) | 1 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 2 | 0
Vulvitis (Infections and infestations) | 1 | 0 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0 | 0
Weight decreased (Investigations) | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other